CLINICAL TRIAL: NCT02884284
Title: Creation of a Prospective and Retrospective Breast Cancer Database
Brief Title: Prospective and Retrospective Breast Cancer Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 15HLSEIN01
Record Dates: First submitted 2016-07-28; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; database
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and tumor samples of patients treated for breast cancer
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: clinical biological database collection

SUMMARY:
In order to accelerate border crossing between basic research and clinical research in breast cancer, it is necessary to easily use clinical and biological data. That is the reason why it is very important to create a clinical, biological and pathologic beast cancer database, mainly prospective but also retrospective. All data are from patients treated in Toulouse Centre.

The scientific community will easily have access to clinical and biological informations through a centralized, structured database , leading to optimize patients with breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Histologically confirmed breast cancer of any stage
* Affiliated to a social security system in france
* Who signed the informed consent

Exclusion Criteria:

* Any psychiatric or medical condition that would make the patient unable to give a signed informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patient with breast cancer of any stage
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-02; Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Database of patients with breast cancer | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Florence DALENC, MD, Principal Investigator — Institut claudius regaud Toulouse ONCOPOLE
Locations (1):
- Institut claudius regaud IUCT ONCOPOLE, Toulouse, France

IPD SHARING:
Plan to Share IPD: No